CLINICAL TRIAL: NCT02305511
Title: A Comparison of Four Intraosseous Access Devices With Standard Venous Catheterization During Child Cardiopulmonary Resuscitation Simulation: a Randomized Crossover Trial.
Brief Title: Intraosseous Access During Pediatric Resuscitation
Acronym: IOCPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IO/2014/01
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
Keywords: Catheterization; Peripheral
MeSH Terms: conditions — Heart Arrest | interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peripheral venous catheterization (Experimental): Peripheral venous catheterization during pediatric resuscitation
  Interventions: Device: Peripheral venous catheterization
- intraosseous access (Experimental): Intraosseus access using intraosseous access devices during resuscitation
  Interventions: Device: Jamshidi; Device: BIG; Device: Cook; Device: EZIO

INTERVENTIONS:
Device: Peripheral venous catheterization — Cannulation using standard method
  Arms: Peripheral venous catheterization
Device: Jamshidi — intraosseous access using the Jamshidi device
  Arms: intraosseous access
Device: BIG — intraosseous access using the BIG device
  Other Names: Bone Injection Gun
  Arms: intraosseous access
Device: Cook — intraosseous access using the Cook device
  Arms: intraosseous access
Device: EZIO — intraosseous access using the EZIO device
  Arms: intraosseous access

SUMMARY:
The purpose of this study was to compare the Jamshidi, the BIG, the Cook, the EZIO intraosseous devices to standard peripheral venous catheterization during pediatric resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel - EMS-paramedics

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Success rate on first attempt | 1 day

SECONDARY OUTCOMES:
Ease of use | 1 day
  Ease of use as reported by participants
Time to successfully perform | 1 day
  Time to successfully perform the intraosseous access

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland